CLINICAL TRIAL: NCT01400620
Title: Phase 2 Study to Evaluate the Safety and Efficacy of IZN-6N4 for the Prevention of Chemo-Radiation-Induced Oral Mucositis in Patients With Head and Neck Cancer
Brief Title: Safety and Efficacy of IZN-6N4 Oral Rinse for the Prevention of Oral Mucositis in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Izun Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IOM-HNC-201-IL
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Oral Mucositis
Keywords: oral mucositis; chemoradiation; head and neck cancer
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active oral rinse (Experimental): Oral rinse containing botanical extracts
  Interventions: Drug: IZN-6N4
- Placebo rinse (Placebo Comparator)
  Interventions: Drug: IZN-6N4

INTERVENTIONS:
Drug: IZN-6N4 — Oral rinse containing 1% botanical extracts, 15 cc rinse 3 times per day, for up to 9 weeks

SUMMARY:
The purpose of this study is to determine whether an oral rinse composed of botanical extracts is effective in the prevention of severe inflammation of the lining of the oral cavity caused by chemotherapy and radiation therapy for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of head and neck cancer
* planned treatment course to include Cisplatin and radiation therapy, cumulative prescription dose between 50-70 Gy
* able to eat at least soft solids
* normal cardiac function
* able to perform oral rinse

Exclusion Criteria:

* Induction chemotherapy regimen
* life threatening allergic reaction to food and/or drugs
* history of any other primary malignancy diagnosed within the past 5 years
* prior radiation to the sites to be treated
* active infections of the oral cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Proportion of WHO score 3-4 Oral Mucositis at a Cumulative Radiation Dosage of 50 Gy in the active and Placebo Groups | Participants will be assessed twice per week during the duration of chemoradiation therapy anticipated to be 5-7 weeks. Following chemoradiation therapy the participants will be assessed weekly for two weeks.
  Degree of oral mucositis will be scored using WHO scoring system bi-weekly throughout course of the trial

SECONDARY OUTCOMES:
Incidence of grade 2-3-4 Oral Mucositis as measured by the WHO scale at increasing increments of cumulative radiation exposure | Participants will be assessed twice per week during the duration of chemoradiation therapy anticipated to be 5-7 weeks. Following chemoradiation therapy the participants will be assessed weekly for two weeks.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (4):
  - UF Health Cancer Center, Gainesville, Florida
  - University of Miami-Sylvester CCC Clinical Research Services, Miami, Florida
  - Mount Sinai Beth Israel - Phillips Ambulatory Care Center, New York, New York
  - NYU Clinical Cancer Center, New York, New York
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Rabin Medical Center - Beilinson Campus, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
  - Assuta Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky